CLINICAL TRIAL: NCT04508348
Title: A Single Center Randomized Controlled Trial to Decrease Length of Stay in Infants With Neonatal Abstinence Syndrome (NAS) With an Exclusive Human Milk Diet
Brief Title: Clinical Trial to Decrease Length of Stay in Infants With Neonatal Abstinence Syndrome With an Exclusive Human Milk Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20200179H
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: human milk
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Milk, Human; Standard of Care

STUDY DESIGN:
Intervention Model Description: A randomized, blinded, controlled trial
Who Masked: Investigator
Masking Description: Physician Investigator will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive Human Milk (Active Comparator): Group One will receive an exclusive human milk diet throughout the 28-day feeding period or until hospital discharge
  Interventions: Other: Human Milk
- Maternal human milk or Formula (Other): Group Two (Control Group) will receive maternal human milk or formula (per standard of care).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Human Milk — Exclusive Human Milk diet
  Other Names: 100% Human Milk
  Arms: Exclusive Human Milk
Other: Standard of Care — This diet will include mother's milk and/or formula
  Other Names: Mother's milk and/or formula
  Arms: Maternal human milk or Formula

SUMMARY:
A clinical trial to evaluate length of stay, growth velocity and clinical outcomes in infants with neonatal abstinence syndrome receiving an exclusive human milk diet. Human milk is defined as expressed human milk or donor milk and its derivatives, human milk-based fortifier and human milk caloric fortifier.

DETAILED DESCRIPTION:
This is a single blinded (physician investigator), randomized, controlled trial to evaluate length of stay in infants with NAS and an exclusive human milk diet during their initial hospitalization after birth and through the 28 days of life or hospital discharge, whichever comes first.

Subjects will be randomized to one of two groups after at birth. Parents who decline participation for their infants in the study will be asked to consent to data gathering on their infants who will be treated and fed per institutional practice. The data on these individuals will be summarized and evaluated descriptively in comparison with the actual trial results.

All experimental group participants will receive exclusive maternal human milk or donor human milk prior to randomization. Once randomized, patients in Group One will receive an exclusive human milk diet throughout the 28-day feeding period or until hospital discharge, whichever comes first. Patients in Group Two (Control Group) will receive maternal human milk or formula (per standard of care). Fortification will be implemented with a standard protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Term infants (≥37 and 0/7 weeks gestational age) ≤ 2 days old with a diagnosis or at risk for neonatal abstinence syndrome. Can be enrolled ante-natally.
2. Infant feeding was NPO (nil per os) or consisted of 100% human milk diet prior to randomization.
3. Parent(s) willing to sign informed consent.
4. Parent(s) willing to comply with study follow-up procedures.

Exclusion Criteria:

1. Term infants >2 days old at the time of evaluation for NAS.
2. <37 weeks gestation.
3. Outborn infants who received enteral nutrition at the other institution prior to transfer. If it is uncertain if infant received even 1 bottle or a small amount of formula, infants will be excluded.
4. Major congenital abnormalities:

   1. Confirmed or suspected major genetic abnormalities (lethal or with extremely low probability for survival).
   2. Chromosomal abnormalities: Trisomies (13, 18, 21 etc.) deletions or translocations (Turner/Williams Syndrome, DiGeorge, to name a few).
   3. Major organ system abnormalities not related to a genetic syndrome that are lethal or have extremely low probability for survival (i.e, bilateral kidney intrinsic disease, pulmonary hypoplasia, CNS (central nervous system) malformations: Arnold Chiari, myelomengoceles, hydranencephaly, squizencephaly, holoprocencephaly).
5. Any comorbidity or significant clinical event prior to enrollment, deemed by the Investigator as likely to affect survival or intestinal health.
6. Legally Authorized Representative(s) unwilling to comply with an exclusive human milk diet either in the form of mother's milk, human milk-based human milk fortifier, human milk based caloric fortifier or donor human milk during the initial hospitalization period and through the 28 day feeding period or hospital discharge, whichever comes first.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | Baseline to 28 days
  Length of stay in infants at risk for neonatal abstinence syndrome who are fed an exclusive human milk diet from birth through the 28-day feeding period or until hospital discharge, whichever comes first

SECONDARY OUTCOMES:
Growth Velocity Rate | Baseline to 28 days
  rate of linear growth and incremental rate of head circumference growth; gm/week, cm/week and z-score from World Health Organization (WHO) growth charts
Body Composition Percentage Fat | 28 days
  Body composition using Peapod at 28 days or discharge. The PEA POD uses the principles of wholebody densitometry to determine body composition. In this technique, body mass and body volume are measured (both performed within the unit). Once body density (Density = Mass/Volume) is determined, the PEA POD uses known (or user customized) densitometric equations to calculate percent Fat.
Body Composition Percentage Fat Free Mass | 28 Days
  Body composition using Peapod. The PEA POD uses the principles of wholebody densitometry to determine body composition. In this technique, body mass and body volume are measured (both performed within the unit). Once body density (Density = Mass/Volume) is determined, the PEA POD uses known (or user customized) densitometric equations to calculate percent Fat-Free Mass.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Blanco, MD, MSCI-TS, Principal Investigator — University of Texas Health at San Antonio
Locations (2):
- United States (2):
  - University Health System, Robert B Green, San Antonio, Texas
  - MARC - The University of Texas Health Science Center, San Antonio, Texas